CLINICAL TRIAL: NCT03003611
Title: Observational Study on the Impact of Hypnose Used as Sedation in the Oncology Surgery in Breast Cancer
Brief Title: Observational Trial on the Impact of Hypnose Used as a Sedation in Oncology Surgery in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: ONCO-GYNECO 2014/1
Record Dates: First submitted 2014-06-19; First posted 2016-12-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2016-12

CONDITIONS: Early Stage Breast Carcinoma
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hypnose: the group of patient who's operated under hypnose sedation
  Interventions: Procedure: hypnose sedation
- traditional anesthesia: The match is realized with a patient operated in the same period as the patient in the hypnose group and it's need a comparative type of surgery.
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: hypnose sedation — Patient will be anesthetized with an hypnose sedation and a complement with light anesthesia
  Groups: Hypnose
Procedure: general anesthesia — Patient will be anesthetized with a classical general anesthesia
  Groups: traditional anesthesia

SUMMARY:
The investigators will compare the operated patients for a beginning breast cancer in the Hypnose arm and the patient in the classical general anesthesia arm. It is a Observational study as we cannot randomized patient, (they need to be compliant with Hypnose).

Patient will be informed that some parameters, about his recovery, will be collected from their medical file. They will not have another particular treatment because they are in the study. It is just a prospective data collection.

The patient will be compared on several items after the surgery ( as pain and pain killer intake, the heal process of the scar, etc...) Also the investigators will compare the impact of hypnose on the other treatments the patient received.

The investigators need approximately 150 patients (Half in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent Form
* In situ breast cancer (early stage)
* Infiltrated Breast cancer (early stage)

Exclusion Criteria:

* No hypnoses is possible for this patient surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient who will benefit of a surgery according a early stage of in-situ or infiltrated breast cancer
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
How is the recovering of the patient according his pain and anxiety, one day after the surgery? Is he anxious; does algique, both or none of the two? Each patient will be categorized according the score they obtain in the different scales. | One day after the surgery
  We'll collect the following information in the standard medical file :
  The collected measures who will analyzed are anxiety, pain and consumption of analgesic.
  Items :
  1. Anxiety (will be mesured by the anxiety visual scale)
  2. Pain (mesured by analogic visual pain scale)
  3. consumption of analgesic (Yes / No - in case o YES : Type, duration, quantity per day) All the responses to the item will be reported and a conclusion between the part of anxiety and the part of the pain will be combine (ex : patient is anxious and have no pain, patient have pain and anxiety, patient have pain and no anxiety, patient have no pain and no anxiety).

SECONDARY OUTCOMES:
How is the recovering of the patient according his pain and anxiety, seven days after the surgery? Is he anxious; does algique, both or none of the two? Each patient will be categorized according the score they obtain in the different scales. | 7 days after surgery
  We'll collect the following information in the standard medical file :
  The collected measures who will analyzed are anxiety, pain and consumption of analgesic.
  Items :
  1. Anxiety (will be mesured by the anxiety visual scale)
  2. Pain (mesured by analogic visual pain scale)
  3. consumption of analgesic (Yes / No - in case o YES : Type, duration, quantity per day) All the responses to the item will be reported and a conclusion between the part of anxiety and the part of the pain will be combine (ex : patient is anxious and have no pain, patient have pain and anxiety, patient have pain and no anxiety, patient have no pain and no anxiety).
Is the quality of the process of cure of the scar normal seven days after the surgery (according that the normal healing process is without infection and hypertrophie)? | 7 days post surgery
  We'll collect the following information in the standard medical file :
  * Redness of the skin : yes /no
  * Delay in the scar process : yes/ no
  * Infection: yes/ no
  * Hypertrophie of the scar : yes/no
  * Pain : Yes/No After analysis of the parameters, we will determine a good scar healing process, or not.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Berlière, MD PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc - UCL, Brussels, Belgium

REFERENCES:
- [Derived] Berliere M, Roelants F, Watremez C, Docquier MA, Piette N, Lamerant S, Megevand V, Van Maanen A, Piette P, Gerday A, Duhoux FP. The advantages of hypnosis intervention on breast cancer surgery and adjuvant therapy. Breast. 2018 Feb;37:114-118. doi: 10.1016/j.breast.2017.10.017. Epub 2017 Nov 11. PMID 29136523